CLINICAL TRIAL: NCT05848011
Title: A Phase 2, Randomized, Open-Label, Study of Lorigerlimab With Docetaxel or Docetaxel Alone in Participants With Metastatic Castration-Resistant Prostate Cancer
Brief Title: A Study of Lorigerlimab With Docetaxel or Docetaxel Alone in Participants With Metastatic Castration-Resistant Prostate Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: MacroGenics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP-MGD019-02
Record Dates: First submitted 2023-04-17; First posted 2023-05-08 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Androgen-Independent Prostatic Cancer; Androgen-Independent Prostatic Neoplasms; Prostate Cancer Recurrent; Androgen-Insensitive Prostatic Cance; Androgen-Resistant Prostatic Cancer; Hormone Refractory Prostatic Cancer; Immunotherapy; Immune Checkpoint Inhibitor; Inhibitory Checkpoint Molecule
MeSH Terms: conditions — Prostatic Neoplasms, Castration-Resistant | interventions — Docetaxel; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Lorigerlimab + Docetaxel and Prednisone (Experimental): Lorigerlimab 6 mg/kg IV (up to 2 years) and docetaxel 75 mg/m^2 IV every 3 weeks (up to 7 months) and prednisone 5 mg orally twice daily (up to 7 months).
  Interventions: Biological: lorigerlimab; Drug: docetaxel; Drug: Prednisone
- Standard of care docetaxel and prednisone (Other): Docetaxel 75 mg/m^2 IV every 3 weeks and prednisone 5 mg orally twice daily.(up to 7 months)
  Interventions: Drug: docetaxel; Drug: Prednisone

INTERVENTIONS:
Biological: lorigerlimab — Lorigerlimab is a DART® molecule that binds PD-1 and CTLA-4
  Other Names: MGD019
  Arms: Lorigerlimab + Docetaxel and Prednisone
Drug: docetaxel — Docetaxel Injection is a cytotoxic anticancer drug approved to treat prostate cancer
  Other Names: Taxotere®
Drug: Prednisone — A corticosteroid drug approved for use with docetaxel in the treatment of prostate cancer

SUMMARY:
The purpose of this study is to determine whether the amount of time before disease progression can be prolonged in participants with metastatic castration-resistant prostate cancer (MCRPC) who receive lorigerlimab in addition to the standard of care (SOC) of docetaxel and prednisone. About 150 participants with mCRPC will be enrolled. Participants will be randomized in a 2:1 ratio to receive lorigerlimab with docetaxel and prednisone (experimental arm) or docetaxel and prednisone alone (standard-of-care arm).

Lorigerlimab+docetaxel or docetaxel will be administered intravenously (IV) in clinic on Day 1 of each 3-week cycle. Prednisone will be administered orally twice daily. Lorigerlimab will be administered for up to 35 cycles. Docetaxel and prednisone will be administered up to 10 cycles until treatment discontinuation criteria are met. Participants will undergo regular testing for signs of disease progression using computed tomography (CT) scans, magnetic resonance imaging (MRI) and prostate-specific antigen (PSA) blood tests. Participants will be asked to complete questionnaires about their health and well-being. Routine examinations and blood tests will be performed and evaluated by the study doctor.

Participants who have disease progression standard-of-care arm have the option of continuing on the study to receive lorigerlimab monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic castration-resistant adenocarcinoma of the prostate without evidence of neuroendocrine differentiation, signet cell, or small cell features.
* Participants must have ≥ 1 metastatic (measurable or non-measurable per PCWG3) lesion.
* Participant has prostate cancer progression at study entry based on PCWG3 criteria.
* Participant shows evidence of disease progression after receiving at least 1 prior androgen receptor axis-targeted therapy (ARAT) regimen (e.g., abiraterone, enzalutamide, apalutamide, or darolutamide).
* Patients with known history of documented breast cancer gene (BRCA) mutation (germline or somatic) must have received an approved poly ADP ribose polymerase (PARP) inhibitor regimen.
* Participants must have adequate performance status, life expectancy and laboratory values.

Exclusion Criteria:

* Any condition preventing participant's ability to receive, tolerate, or comply with the planned treatment or study procedures.
* Received prior chemotherapy for mCRPC or checkpoint inhibitors for prostate cancer.
* Current active or chronic infections.
* Any clinically significant heart, lung, or gastrointestinal disorders.
* Allergy to any of the study treatments or components of the study treatments.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2023-09-28 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Median radiographic progression free survival (rPFS) determined by investigator review. | Every 9 weeks for the first year, followed by every 12 weeks for up to 3 more years
  The rPFS is defined as the time from the date of randomization to the date of first documented PD per Prostate Cancer Working Group 3 (PCWG3) criteria or death from any cause, whichever occurs first.

SECONDARY OUTCOMES:
Objective response rate (ORR) per PCWG3 criteria | Every 9 weeks for the first year, followed by every 12 weeks for up to 3 more years
  ORR is defined as the number of participants who have a best overall response of confirmed complete response (CR) or partial response (PR) without prior confirmed bone progression
Duration of response (DoR) | Every 9 weeks for the first year, then every 12 weeks for up to 4 years
  DoR is the time from the date of initial tumor response (CR or PR) to the date of first disease progression or death from any cause, whichever occurs first.
Time to response (TTR) | Every 9 weeks for the first year, followed by every 12 weeks for up to 3 more years
  TTR is defined as the time from the start of treatment to the first objective response (CR or PR).
PSA50 response rate | Every 3 weeks up to 2 years, followed by every 12 weeks for up to 2 more years
  PSA50 response is defined as a ≥ 50% decline in PSA from baseline with confirmation at least 3 weeks after the first documented reduction in PSA of ≥ 50%.
PSA90 response rate | Every 3 weeks up to 2 years, followed by every 12 weeks for up to 2 more years
  PSA90 response is defined as a ≥ 90% decline in PSA from baseline with confirmation at least 3 weeks after the first documented reduction in PSA of ≥ 90%.
Time to PSA progression | Every 9 weeks for the first year, followed by every 12 weeks for up to 2 more years
  Time to PSA progression is defined as the time from the date of randomization to the first documented PSA progression.
Duration of PSA response | Every 3 weeks up to 2 years, followed by every 23 weeks for up to 2 more years.
  Duration of PSA response is defined as the time from the date of first PSA response to the earliest date of PSA progression.
Overall survival (OS) | Throughout the study up to 4 years
  OS is defined as the time from the date of randomization to the date of death from any cause.
Time to First Symptomatic Skeletal Event (SSE) | Throughout the study up to 4 years
  Time to first SSE is defined as the time from the date of randomization to the first occurrence of SSE from any cause.
Time to pain progression using the BPI-sf questionnaire | Every 9 weeks for the first year, followed by every 12 weeks for up to 2 more years
  Time to pain progression is defined as the time interval from randomization to the first date a participant experiences pain progression. Higher scores indicate more severe pain.
Pain severity using the Brief Pain Index - short form (BPI-sf) questionnaire | Every 3 weeks up to 2 years
  The BPI-sf pain severity score consists of 4 items that assess pain at its worst, least, average, and current pain intensity. The pain severity score is the average of the 4 item scores. Higher scores indicate more severe pain.
Pain interference using the BPI-sf questionnaire | Every 3 weeks up to 2 years
  The BPI-sf pain interference score includes 7 items: general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life. The pain interference score is the average of the 7 interference items. Higher scores indicate more interference from pain in daily life.
Functional Assessment of Cancer Therapy-Prostate (FACT-P) questionnaire | Every 3 weeks up to 2 years
  The FACT-P consists of 27 items from the Functional Assessment of Cancer Therapy-General (FACT-G) that measure physical, social/family, emotional, and functional well-being and 12 items that compose the Prostate Cancer Subscale (PCS). Higher scores indicate greater impact of prostate cancer on daily life.
Description of types of adverse events (AEs) between treatment groups. | Throughout treatment up to 27 months
  Number of participants with adverse events (AEs), serious adverse events (SAEs), and AEs leading to study treatment discontinuation
Lorigerlimab maximum concentration or concentration at the end of infusion (Cmax) | Every 21-day cycle throughout the study, for an average of 1 year.
  The highest measured concentration of lorigerlimab in the bloodstream.
Lorigerlimab area under the concentration time curve (AUC) | Every 21-day cycle throughout the study, for an average of 1 year.
  AUC is the total amount of lorigerlimab in bloodstream after drug administration
Trough drug concentration (Ctrough or Cmin) | Every 21-day cycle throughout the study, for an average of 1 year.
  Trough concentration is the concentration measured before a subsequent dose of lorigerlimab
Clearance (CL) | Every 21-day cycle throughout the study, for an average of 1 year.
  Drug clearance is the amount of drug removed from the bloodstream by the body per unit of time
Volume of distribution (Vz) | Every 21-day cycle throughout the study, for an average of 1 year.
  The volume of distribution is related to how much drug is distributed to body tissues, or remains in the bloodstream.
Terminal half-life | Every 21-day cycle throughout the study, for an average of 1 year.
  Terminal elimination half-life is the time it takes for the concentration of the drug in plasma or serum to be reduced by 50%
Number of participants who develop anti-drug antibodies | Throughout the study, up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Denise Casey, M.D., Study Director — MacroGenics
Locations (49):
- United States (6):
  - United Medical Group, Miami, Florida
  - Orlando Health Cancer Institute, Orlando, Florida
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Nebraska Cancer Specialists, Grand Island, Nebraska
  - MD Anderson Cancer Center, Houston, Texas
  - University of Virginia Health System Cancer Center, Charlottesville, Virginia
- Australia (3):
  - Peter MacCallum Cancer Centre, North Melbourne
  - North Shore Private Hospital, St Leonards
  - Westmead Hospital, Westmead
- Belgium (3):
  - Cliniques universitaires Saint-Luc (CUSL), Brussels, Brussels
  - UZ GENT, Ghent
  - Centre Hospital de l'Ardenne, Libramont
- Bulgaria (2):
  - Comprehensive Cancer Center, Plovdiv
  - UMHAT Sv. Ivan Rilski, Sofia
- France (9):
  - Institut Bergonie, Bordeaux
  - Clinique Victor Hugo, Le Mans
  - Centre Léon Bérard, Lyon
  - Centre Antoine Lacassagne, Nice
  - Institut Mutualiste Montsouris, Paris
  - Centre Hospitalier Quimper, Quimper
  - CHP Saint Grégoire, Saint-Grégoire
  - Hia Begin, Saint-Mandé
  - Hopital Foch, Suresnes
- Georgia (8):
  - LTD High Tech Hosp Medcenter, Batumi
  - First University Clinic TSMU, Tbilisi
  - LTD Consilium Medulla, Tbilisi
  - Ltd Gidmedi, Tbilisi
  - LtD L.M.National Urology Center, Tbilisi
  - LTD MMT Hospital, Tbilisi
  - LTD Todua Clinic, Tbilisi
  - Onc. Scient. Research Center, Tbilisi
- Poland (4):
  - Przychodnia Lekarska KOMED, Konin
  - Pratia McM Kraków, Krakow
  - Europejskie Centrum Zdrowia Otwock, Szpital im. Fryderyka Chopina, Otwock
  - Szpital Grochowski im. dr med. Rafała Masztaka Sp. z o.o., Oddział Chemioterapii, Warsaw
- Pan American Center for Oncology Trials, LLC, Rio Piedras, Puerto Rico
- Spain (9):
  - H U Germans Tries i Pujol, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Sant Pau, Barcelona
  - Institut Català d'Oncologia Hospitalet_ICO Hospitalet, Barcelona
  - Vall d' Hebron Institute of Oncology (VHIO), Barcelona
  - Hospital 12 de octubre, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
  - FIVO: Instituto Valenciano de Oncología, Valencia
- United Kingdom (4):
  - Churchill Hospital, Headington
  - Charing Cross Hospital, London
  - Royal Marsden Hospital, Sutton
  - Musgrove Park Hospital, Taunton

IPD SHARING:
Plan to Share IPD: No